CLINICAL TRIAL: NCT01000948
Title: An Open Phase II, Two-centre, 1-Arm Safety Study of Once-daily Orally Administered 10 mg ZD4054 in Prior Chemotherapy Treated Patients With Metastatic Hormone-resistant Prostate Cancer
Brief Title: A Safety Study of ZD4054 in Prior Chemotherapy Treated Patients With Metastatic Hormone-resistant Prostate Cancer
Acronym: DAPROCA-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A consequence of the results of the ENTHUSE phase III study program
Sponsor: Aarhus University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Borre, Professor, DMSci, PhD, Aarhus University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISSIS40540005; DAPROCA-1
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2011-07

CONDITIONS: Prostate Cancer; Metastasis
Keywords: Prostate cancer; Castration resistant; Chemotherapy resistant; Endothelial receptor A inhibitor; ZD4054
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZD4054 (Experimental): The study had only one arm: intervention
  Interventions: Drug: ZD4054

INTERVENTIONS:
Drug: ZD4054 — ZD4054 10 mg given orally, once daily in tablet form to all patients in two years or until investigator consider the drug for useless.

SUMMARY:
This is a prospective, open, one-arm, two-centre, Phase II clinical safety pilot-study. The trial is designed to gain initial safety and efficacy-related data on once-daily orally administered ZD4054 10 mg in prior chemotherapy treated patients with metastatic hormone-resistant prostate cancer.

DETAILED DESCRIPTION:
Study centres and number of patients planned This pilot study will be conducted in approximately 24 patients recruited from two hospital-based Danish centres: department of Urology K, Aarhus University Hospital, Skejby and department of Urologic Surgery D, Rigshospitalet. The recruitment of patients will be competitive among centres. 1-2 months before expected LSI it should be discussed if the target accrual should be expanded.

Study period Phase of development Estimated date of first patient enrolled August 1th 2009 II Estimated date of last patient completed July 31th 2012 Total study duration is approximately 36 months, which includes 12 months' recruitment, 36-month follow-up for safety and final survival analysis.

Objectives

The primary objective of this study is:

To assess the safety and tolerability profile of ZD4054 after treatment with chemotherapy

* Adverse events
* Vital signs
* Laboratory data
* ECGs
* Physical Exam
* Death from any cause

The secondary objectives of the study are:

1. To investigate the effect of ZD4054 on rate of rise of PSA
2. To investigate the effect of ZD4054 on prostate cancer related pain
3. To investigate the effect of ZD4054 on the plasma concentration of circulating tumour cells (CTC).

In addition, Time to Progression and Overall Survival (time to death) will be compared with historical data in a post chemotherapy population.

Study design This is a prospective, Open, One-arm, Phase II clinical safety pilot-study. The trial is designed to gain initial safety and efficacy-related data on once-daily orally administered ZD4054 10 mg in prior chemotherapy treated patients with metastatic hormone-resistant prostate cancer.

Patients could receive other therapies including prednisolone, estramustine, ketoconazole and second-line or third-line antiandrogens at investigator's discretion without being considered treatment failures or having to stop study therapy; however every attempt will be made to avoid changes in medication for at least 12 weeks to minimise potential for confounding on study endpoints over this time period. Chemotherapy and radiation therapy may also be administered in addition to study therapy at investigator's discretion after objective progression if the patient is considered likely to derive benefit. Patients will be followed to death.

Target patient population A total number of 24 male patients aged 18 years or older with metastatic hormone-resistant prostate cancer who have progressive disease (defined by rising serum prostate-specific antigen levels despite medical or surgical castration) and previously received cytotoxic chemotherapy (docetaxel) for the treatment of HRPC.

Investigational product, dosage and mode of administration

Patients will not be randomised and all patients will receive:

• ZD4054 10 mg given orally, once daily in tablet form. Duration of treatment Patients will receive daily ZD4054 as long as they meet no withdrawal criteria. Following completion of 24 months of ZD4054, patients, who in the investigator's opinion are experiencing benefit from study treatment, may continue on ZD4054, for as long as they meet no withdrawal criteria.

Statistical methods The study is a pilot study designed to collect safety/tolerability data and assess markers of efficacy. A total of 24 patients will be recruited into this pilot study and this is based primarily on the number of patients that can be recruited in a reasonable time period at the centres and should be sufficient to make an initial assessment of safety/tolerability and the efficacy markers.

For the assessment of tolerability and safety, incidence and severity of adverse events (AEs) (based on National Cancer Institute Common Terminology Criteria for Adverse Events, version 3 (NCI CTCAE) grading), laboratory values, vital signs, ECGs and physical exam will be summarised.

Secondary endpoints will be presented and analysed to investigate trends in the data. The interpretation of the analyses will consider the number of assessments being undertaken.

Pain will be assessed using the Brief Pain Inventory Demography and baseline data will be summarised. Any analyses will be performed using SPSS and other validated software as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Male, aged 18 years or older
3. Histological or cytological confirmation of adenocarcinoma of the prostate
4. Documented evidence of bone metastasis on bone scans.
5. Surgically castrated or continuously medically castrated with serum testosterone less than 2.4 nmol/L (70 ng/dL).
6. Previously (not inside 8 weeks) treated with at least two times 75 mg/m2 docetaxel.
7. Biochemical progression of prostate cancer after chemotherapy, documented while the patient is castrate:

   o Biochemical progression is defined as at least 2 stepwise increases (≥1ng/mL) in PSA over a period of ≥1 month (values do not need to be consecutive but 2 values that have increased since the previous highest value are required) with at least 14 days between each measurement irrespective of assay or laboratory.
8. Life expectancy of 3 months or more.

Exclusion Criteria:

1. Use of potent CYP450 inducers (such as phenytoin, rifampicin, carbamazepine, phenobarbitone and St John's Wort) within 2 weeks of starting study treatment. Dexamethasone will be allowed if the investigator feels it is necessary but is encouraged to use a different form of steroid treatment wherever possible
2. Have received investigational drug in another clinical study of anticancer therapy, within 4 weeks of starting study treatment
3. Hypersensitivity to endothelin antagonists
4. Neurological symptoms or signs consistent with acute or evolving spinal cord compression. If a patient has neurologic symptoms, an MRI must be performed that demonstrates no impending or actual spinal cord compression. Stable, previously treated patients are allowed
5. History of past or current epilepsy, epilepsy syndrome, or other seizure disorder
6. Stage II, III or IV cardiac failure (classified according to New York Heart Association (NYHA) classification) or myocardial infarction within 6 months prior to study entry
7. QT interval corrected for heart rate e.g., by Bazett's correction >470 msec
8. In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease (e.g., currently unstable or uncompensated respiratory, cardiac, hepatic or renal disease) or evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
9. Hemoglobin (Hb) <5 mmol/L. Concomitant use of erythropoietin or blood transfusions is allowed
10. Serum bilirubin >1.5 times the upper limit of normal (ULN). This will not apply to patients with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of haemolysis or hepatic pathology), who will be allowed in consultation with their physician
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 times the ULN or 5 times the ULN in the presence of liver metastasis
12. Creatinine clearance of <50 mL/minute, determined using the Cockcroft-Gault equation or by 24-hour creatinine clearance

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability profile of ZD4054 after treatment with chemotherapy | 2 years
Adverse events | 2 years
Vital signs | 2 years
Laboratory data | 2 years
ECGs | 2 years
Physical Exam | 2 years
Death from any cause | 2 years

SECONDARY OUTCOMES:
To investigate the effect of ZD4054 on rate of rise of PSA | 2 years
To investigate the effect of ZD4054 on prostate cancer related pain | 2 years
To investigate the effect of ZD4054 on the plasma concentration of circulating tumour cells (CTC). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borre, MD Phd DMSc, Study Chair — Dpt Urology Aarhus University Hospital - DAPROCA
Locations (1):
- Dpt of Urology,Aarhus University Hospital, Aarhus, Denmark